CLINICAL TRIAL: NCT03190733
Title: A Randomized,Open,Multicenter and Prospective Study of the Optimized Dose of Anti-Thymoglobuline in Haploidentical Allogeneic Stem Cell Transplantation
Brief Title: A Optimal Anti-Thymoglobuline (ATG) Dose Decrease cGVHD But Not Increase Leukemia Relapse for Haplo-HSCT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhujiang Hospital (Other)
Collaborators: Nanfang Hospital, Southern Medical University (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); Second Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2016-XYNK-001
Record Dates: First submitted 2017-06-15; First posted 2017-06-19 (Actual); Last update posted 2017-06-19 (Actual); Status verified 2016-12

CONDITIONS: Chronic Graft-versus-host-disease; Leukemia Relapse
Keywords: Hematopoietic Stem Cell Transplantation; ATG; chronic GVHD; leukemia relapse
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — fludarabine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ATG 10.0mg/kg (Experimental): ATG 10.0mg/kg group refers to treatment with ATG in the total dose of 10.0mg/kg.
  Interventions: Drug: ATG
- ATG 12.5mg/kg (Active Comparator): ATG 12.5mg/kg group refers to treatment with ATG in the total dose of 12.5mg/kg.
  Interventions: Drug: ATG

INTERVENTIONS:
Drug: ATG — ATG will be intravenously infused via a central venous catheter in 4 or 5 days, from day -4 or -3 until day 0. The other conditioning drugs administered before transplantation include fludarabine (Flu), busulfan (Bu),cyclophosphamide (Cy). All transplant recipients will receive cyclosporine A (CsA), mycophenolate mofetil(MMF) for aGVHD prevention.
  Other Names: fludarabine

SUMMARY:
In this study, a randomized, prospective, multicenter, open cohort study was conducted to investigate patients with acute leukemia (14～60-year-old) with different ATG doses (10 mg / kg and 12.5 mg / kg ) in fludarabine, busulfan, cyclophosphamide and antilymphocyte globulin (FBCA) pretreatment protocol of Haploidentical hematopoietic stem cell transplantation (haplo-HSCT). The purpose is to compare the incidences of chronic graft vs host disease (cGVHD) in haplo-HSCT recipients receiving different dose ATG and one year leukemia relapse after transplantation. The main objective was to investigate the optimal dose of ATG for decrease cGVHD and not increase one year relapse leukemia after haplo-HSCT. Its significance is to provide evidence-based medical evidence to reduce the occurrence of cGVHD and to improve the quality of life of patients with haplo-HSCT.

DETAILED DESCRIPTION:
Human leukocyte antigen (HLA) haploidentical hematopoietic stem cell transplantation is an effective method for the treatment of hematological malignancies. However, high incidence rate of graft-versus-host disease (GVHD) seriously affects the quality of life of patients.

Using ATG in vivo T cell transplantation regimens reduce the rate of acute GVHD (aGVHD) and cGVHD. However, the optimal dose of ATG is unknown, Huang's reported that a prospective, randomized trial, which compared the long-term outcomes of 2 ATG doses used in myeloablative conditioning before unmanipulated haplo-HSCT. Patients were received 10 mg/kg or 6 mg/kg of ATG in conditioning regimen. The 5-year cumulative incidence of cGVHD was found to be higher with ATG 6mg/kg (75.0% vs 56.3% [P = .007] and moderate-to-severe cGVHD: 56.3% vs 30.4% [P<.0001]. ATG 10mg/kg in conditioning regimen was found to be associated with a lower risk of cGVHD. But the moderate-to-severe cGVHD was as high as 35%. We established the FBCA pretreatment regimen which added ATG and achieve the goal of reducing GVHD. In this FBCA pretreatment regimen the ATG dose was 12.5mg/kg which higher than that of other protocol. The cumulative incidence of grades II-IV aGVHD and cGVHD was 21.9% and 14.3% with the 12.5mg/kg ATG in the FBCA conditioning regimen which was lower than that of ATG 10mg/kg reported by Huang. However, ATG may lead to immunosuppression and lead to slow recovery of immune function and increased infection rate and may increase leukemia relapse after transplantation. What is the optimal does of ATG in FBCA pretreatment regimen which could reduce cGVHD and not increase leukemia relapse after transplantation? Access to ClinicalTrials and other sites found that there was still no related international studies with the FBCA conditioning regimen. We hypothesize that total ATG dose 12.5mg/kg in FBCA pretreatment regimen will decrease cGVHD and not increase leukemia relapse post transplantation.

In this study, a randomized, prospective, multicenter, open cohort study was conducted to investigate patients (14～60-year-old) with different ATG doses (10 mg / kg and 12.5 mg / kg ) in the FBCA pretreatment protocol of haploidentical hematopoietic stem cell transplantation. The purpose of this study is to compare the incidences of cGVHD and one year leukemia relapse in haploidentical hematopoietic stem cell transplant recipients receiving different dose of antithymocyte globulin (ATG) for acute graft-versus-host disease(aGVHD) prophylaxis The first objective was to investigate the optimal dose of ATG for decrease cGVHD and not increase one year relapse leukemia after haplo-HSCT. Its significance is to provide evidence-based medical evidence to reduce the occurrence of cGVHD and to improve the quality of life of patients with HLA haploid hematopoietic stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. patients age between 14 yeas old and 60 years old
2. patients with acute myeloid leukemia and acute lymphoblastic leukemia who needed stem cell transplantation without available HLA-identical related or unrelated donors

Exclusion Criteria:

1. Patients with severe infections
2. patients with major organ abnormal including renal, liver, lung or heart.
3. Patients with any conditions not suitable for the trial (investigators' decision)
4. patients age below 14 years old and more than 60 years old.

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 192 (Estimated)
Dates: Start 2017-08-30 (Estimated); Primary Completion 2020-09-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
occurrence of chronic GVHD | from the day of stem cell transplantation to one year after stem cell transplantation
  chronic GVHD diagnosis based on National Institutes of Health (NIH) criterion

SECONDARY OUTCOMES:
one year cumulative incidence of leukemia relapse | from the day of stem cell transplantation to one year after stem cell transplantation
  leukemia relapse base on morphology criterion
The cumulative incidence rate of acute GVHD | from the day of stem cell transplantation to one year after stem cell transplantation
  acute GVHD diagnosis based on NIH criterion
no relapse mortality one year | from the day of stem cell transplantation to one year after stem cell transplantation
  no relapse death

CONTACTS AND LOCATIONS:
Overall Officials: Bingyi Wu, MD, Principal Investigator — Zhejiang Hospital of southern Medical Unversity

IPD SHARING:
Plan to Share IPD: Yes
individual participant data are to be shared with other researchers, when it will be available and be obtained by web.

REFERENCES:
- [Background] Lin X, Lu ZG, Song CY, Huang YX, Guo KY, Deng L, Tu SF, He YZ, Xu JH, Long H, Wu BY. Long-term outcome of HLA-haploidentical hematopoietic stem cell transplantation without in vitro T-cell depletion based on an FBCA conditioning regimen for hematologic malignancies. Bone Marrow Transplant. 2015 Aug;50(8):1092-7. doi: 10.1038/bmt.2015.108. Epub 2015 May 11. PMID 25961770
- [Background] Long H, Lu ZG, Song CY, Huang YX, Xu JH, Xu JX, Deng L, Tu SF, He YZ, Lin X, Guo KY, Wu BY. Long-term outcomes of HLA-haploidentical stem cell transplantation based on an FBCA conditioning regimen compared with those of HLA-identical sibling stem cell transplantation for haematologic malignancies. Bone Marrow Transplant. 2016 Nov;51(11):1470-1475. doi: 10.1038/bmt.2016.170. Epub 2016 Jun 20. PMID 27322852
- [Background] Chang YJ, Wang Y, Mo XD, Zhang XH, Xu LP, Yan CH, Chen H, Chen YH, Chen Y, Han W, Wang FR, Wang JZ, Liu KY, Huang XJ. Optimal dose of rabbit thymoglobulin in conditioning regimens for unmanipulated, haploidentical, hematopoietic stem cell transplantation: Long-term outcomes of a prospective randomized trial. Cancer. 2017 Aug 1;123(15):2881-2892. doi: 10.1002/cncr.30540. Epub 2017 Mar 16. PMID 28301690